CLINICAL TRIAL: NCT02470117
Title: Comparison of the Efficacy of Alginate-based Reflux Suppressant and Magnesium-aluminium Antacid Gel for Treatment of Heartburn in Pregnancy : A Randomized Double-Blind Controlled Trial
Brief Title: Alginate-based Reflux Suppressant and Magnesium-aluminium Antacid Gel for Treatment of Heartburn in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Prof. Vorapong Phupong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 567/57
Record Dates: First submitted 2015-06-05; First posted 2015-06-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Heartburn in Pregnancy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alginate-based reflux suppressant (Active Comparator): Alginate-based reflux suppressant 15 ml oral every 6 hours for 2 weeks
  Interventions: Drug: Alginate-based reflux suppressant
- magnesium-aluminium antacid gel (Sham Comparator): magnesium-aluminium antacid gel 15 ml oral every 6 hours for 2 weeks
  Interventions: Drug: magnesium-aluminium antacid gel

INTERVENTIONS:
Drug: Alginate-based reflux suppressant
  Arms: Alginate-based reflux suppressant
Drug: magnesium-aluminium antacid gel
  Arms: magnesium-aluminium antacid gel

SUMMARY:
This study evaluates the efficacy of alginate-based reflux suppressant and magnesium-aluminium antacid gel for treatment of heartburn in pregnancy. Half of the participants will receive alginate-based reflux suppressant, while the other half will receive magnesium-aluminium antacid gel.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women gestational age less than 36 weeks with heartburn

Exclusion Criteria:

* Having medical disease that contraindicated to use study drug
* Allergic to alginate-based reflux suppressant and magnesium-aluminium antacid gel

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of heartburn as measured by diary chart | 2 weeks

SECONDARY OUTCOMES:
Intensity of hearburn as measured by visual analog scale | 2 weeks
satisfaction as measured by questionnaire | 2 weeks
quality of life as measured by questionnaire SF-8 | 2 weeks
Number of participants with side effects | 2 weeks
fetal outcomes as measured by birth weight and Apgar scores | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University
Locations (1):
- Vorapong Phupong, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Hampson FC, Farndale A, Strugala V, Sykes J, Jolliffe IG, Dettmar PW. Alginate rafts and their characterisation. Int J Pharm. 2005 Apr 27;294(1-2):137-47. doi: 10.1016/j.ijpharm.2005.01.036. PMID 15814238
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Mahadevan U, Kane S. American gastroenterological association institute technical review on the use of gastrointestinal medications in pregnancy. Gastroenterology. 2006 Jul;131(1):283-311. doi: 10.1053/j.gastro.2006.04.049. PMID 16831611
- [Background] Malmud LS, Charkes ND, Littlefield J, Reilley J, Stern H, Rosenberg R, Fisher RS. The mode of action alginic acid compound in the reduction of gastroesophageal reflux. J Nucl Med. 1979 Oct;20(10):1023-8. PMID 231639
- [Background] Richter JE. Review article: the management of heartburn in pregnancy. Aliment Pharmacol Ther. 2005 Nov 1;22(9):749-57. doi: 10.1111/j.1365-2036.2005.02654.x. PMID 16225482
- [Result] Quartarone G. Gastroesophageal reflux in pregnancy: a systematic review on the benefit of raft forming agents. Minerva Ginecol. 2013 Oct;65(5):541-9. PMID 24096290
- [Result] Strugala V, Bassin J, Swales VS, Lindow SW, Dettmar PW, Thomas EC. Assessment of the Safety and Efficacy of a Raft-Forming Alginate Reflux Suppressant (Liquid Gaviscon) for the Treatment of Heartburn during Pregnancy. ISRN Obstet Gynecol. 2012;2012:481870. doi: 10.5402/2012/481870. Epub 2012 Nov 4. PMID 23209926